CLINICAL TRIAL: NCT05273151
Title: An Open Pilot Study to Evaluate the Efficacy of Intranasal Kinetic Oscillation Stimulation in the Preventive Treatment of Chronic Migraine on Patients Not Responding to a Preventive Treatment Targeting the CGRP Pathway
Brief Title: A Study With Intranasal Kinetic Oscillation Stimulation (KOS) in the Prevention of Chronic Migraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusion due to new treatment (Gepants)
Sponsor: Chordate Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PM009
Record Dates: First submitted 2022-01-31; First posted 2022-03-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Intervention Model Description: Open label Investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KOS treatment (Other): Treatment with intranasal kinetic oscillation stimulation (KOS)
  Interventions: Device: KOS (Intranasal kinetic oscillation stimulation)

INTERVENTIONS:
Device: KOS (Intranasal kinetic oscillation stimulation) — Treatment is 10 minutes in each nasal cavity. Totally 2 x 10 minutes per treatment.

SUMMARY:
An open pilot study, non-controlled, single center investigation.

DETAILED DESCRIPTION:
An open pilot study, non-controlled, single center investigation. The study consists of a 4-week screening period, a 6-week treatment period, and a 12 week follow-up period.

Subjects who provided written informed consent and are eligible for the study will be asked to complete a daily diary for 4 weeks during the screening period. In the diary the subjects will record headache and migraine days, any changes in their health, and concomitant medications they may be using. The data collected in the diary during this screening period will be used as Baseline for the performance assessments.

Subjects who completed the screening period and continue to meet the eligibility criteria after review of diary entries by the investigator will receive treatment. The subjects will receive 6 treatments with the Chordate System S220 at weekly intervals at the site (Day 0 to 35; treatment Visit [V] 1 to 6) and continue to maintain a daily diary.

After completion of the 6-week study treatment period (V1 to V6), subjects will be treated monthly and followed up for another 12 weeks. The final visit will be performed on Day 125, 12 weeks after the last study treatment. During the 12-week follow-up, the subjects will continue to complete a daily diary.

ELIGIBILITY:
Inclusion Criteria

1. The subject is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the informed consent form.
2. Male or female aged between 18 and 70 years (inclusive) at the time of providing informed consent.
3. Diagnosed as suffering from chronic migraine with or without aura (≥15 headache days per month including at least 8 migraine days for more than 3 months before screening) according to the International Headache Society classification (International Classification of Headache Disorders III);
4. Migraine onset before the age of 50 years.
5. Reported history of migraine for at least 1 year before screening.
6. If subjects are on a preventive treatment at the time of screening, this must have been stable over the preceding 3 months.
7. If subjects are on preventive treatment at the time of screening, they have to be able and willing to maintain current preventive treatment regimen (no change in type, frequency or dose) from screening to end of follow-
8. Failed at least 3 different preventive medications and 3 months of treatment with a CGRP targeting therapy.
9. Women of childbearing potential must be willing to use highly effective contraceptive methods (failure rate <1% per year when used consistently and correctly) during the study.

Exclusion Criteria

1. Unable to distinguish between migraine and other headache types.
2. An ongoing upper respiratory infection, nasal tumors, or wounds in the nasal cavity.
3. Nasal cavity abnormalities that prevents catheter insertion.
4. A concomitant condition that could cause excessive nose bleeding or ongoing treatment with anticoagulant medication (except Aspirin and Clopidogrel).
5. A known allergy to polyurethane (polyurethane is used in the catheter balloon).
6. Systemic diseases with manifestations in the nose.
7. Previous treatment with radiation therapy to the nasal area.
8. Nasal surgery performed within the last six months.
9. Concurrent condition or risk of non-compliance that, in the investigator's opinion, may affect the interpretation of performance or safety data or which otherwise contraindicates participation in a clinical investigation;
10. Pregnant and lactating women;
11. Participation in a clinical investigation within 3 months of enrolment or planned participation at any time during this clinical investigation;
12. Previous participation in this study;
13. Employees of the study site or the sponsor directly involved with the conduct of the study, or immediate family members of any such individuals;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Mean change in headache days | baseline to 6 weeks
  Change in headache days with moderate to severe intensity after 6 weeks of treatment. Headache days are collected in eDiary

SECONDARY OUTCOMES:
Mean change in Migraine days Mean change of migraine days, responder rate, use of abortive medication, health-related quality of life and disability, and patient's global impression of severity 12 weeks (90 days) | Baseline to 12 weeks
  Migraine days is collected in an eDiary.
Incidence of adverse events (AEs) and adverse device effects (ADEs) | Baseline to 12 weeks
  All adverse events (AEs) and adverse device effects (ADEs) incidence and severity following treatment with the Chordate System 220
Number of patients who are responders | baseline to 12 weeks
  Responders are classified as responder (less migraine/headache days) or non-responder (same or worsening of migraine/headache days).
  A respondes is a patient who has decrease of headaches/migraine days whilst a non responder had no or the same number of headache/migraine days
Number of patients who decrease use of abortive medication | baseline to 12 weeks
  Intake of abortive medications are registred in eDiary and will be calculated on patient level
Mean change in Hospital Anxiety and Depression Scale (HADS) | baseline to 12 weeks
  HADS is a scale with 7 questions related to anxiety and 7 questions related to depression Anxiety can have 0-21 points (lower score means no anxiety) and Depression 0-21 points (higher score means no depression)
Mean change in Headache Impact Test (HIT-6) | baseline to 12 weeks
  HIT-6 consist of 6 questions HIT-6 with scores from 6 to 13 where 13 is worst case per question so lower score means less problems
Mean change in Subject global severity | baseline to 12 weeks
  Patient Global severity is a scale with four (4) scores, where normal (0) is the lowest and show no problems whilst severe (3) is the worst score 0=Normal
  1. Mild
  2. Moderate
  3. Severe
Mean change in headache days | week 6-12
  Change in headache days with moderate to severe intensity from eDiary

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Goadsby, Prof,MD, PhD, Principal Investigator — Wellcome Foundation Building, Denmark Hill Campus King's College London
Locations (2):
- United Kingdom (2):
  - Hull Royal Infirmary, Hull University Teaching Hospital, Hull
  - Wolfson Centre for Age-Related Diseases Institute of Psychiatry, Psychology and Neuroscience Wellcome Foundation Building, Denmark Hill Campus King's College, London

IPD SHARING:
Plan to Share IPD: No
Due to uncertainties in EU data protection legislation individual deidentified participant data are not shared. The main uncertainty is the concept of what "deidentified" means. It appears not to mean that the data set of a person is simply separated from the person's name. What additional operations have to be done appears to depend on technological capabilities to re-identify the persons associated with the data set. A common perception is that the technological capabilities for re-identification are permanently increasing. This could have the effect that public data sets that are regarded as deidentified now might become re-identifiable data sets in the future. Once this happens, the sponsor is no longer able to make the publication of the data sets un-happen. This could result in punishment by EU data protection authorities. The sponsor wants to avoid this.